CLINICAL TRIAL: NCT04167774
Title: Efficacy and Safety of Camrelizumab Combined With Nb-Paclitaxel in Patients With Recurrent/Metastatic Non-small-cell Lung Cancer After the Failure of Platinum-based Therapy
Brief Title: A Study to Evaluate Camrelizumab in Combination With Nb-Paclitaxel in Patients With Advanced or Metastatic NSCLC
Acronym: Compass-001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiuyu Cai, Xiuyu Cai，Principal investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Compass-001
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Immune Checkpoint Inhibitor; nb-Paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; Injections; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab +nb-Paclitaxel (Experimental): Participants receive Camrelizumab 200mg(3mg/kg for underweight patients) iv and nb-Paclitaxel 260mg/m2 iv every 3 weeks until disease progression or unacceptable toxicity
  Interventions: Drug: Camrelizumab; Drug: nb-Paclitaxel

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab will be administered as a 30-minute IV infusion Q3W at a dose of 200mg (3mg/kg for underweight patients).
  Other Names: Camrelizumab for Injection
Drug: nb-Paclitaxel — nb-Paclitaxel will be administered as a 30-minute IV infusion Q3W at a dose of 260mg/m2 for 4-6 cycles.
  Other Names: Paclitaxel for Injection(Albumin Bound)

SUMMARY:
The purpose of this study is to explore the efficacy and safety of Camrelizumab in combination with nb-Paclitaxel in treating patients with recurrent/metastatic non-small-cell lung cancer.

DETAILED DESCRIPTION:
Camrelizumab is a humanized monoclonal antibody against Programmed death 1(PD-1). Albumin-bound paclitaxel is a new nano-paclitaxel drug coated with human albumin. Patients with recurrent/metastatic non-small-cell lung cancer after the failure of platinum-based therapy will received Camrelizumab 200mg((3mg/kg for underweight patients) iv and nb-Paclitaxel 260mg/m2 iv every 3 weeks. The efficacy and safety will be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female ≥ 18 years of age
2. Subjects enrolled must have histologically-confirmed or cytologically confirmed diagnosis of stage ⅢB,Ⅳnon-small cell lung cancer（NSCLC）,at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST)
3. Disease progression experienced during or after one prior platinum containing doublet chemotherapy（excluding taxane chemotherapy）
4. Subjects must have had no more than one prior systemic chemotherapeutic regimen Note: a. Replacement of platinum drugs for toxicity is considered as a systemic chemotherapeutic regimen; b.Subjects with recurrent disease > 6 months after Postoperative adjuvant platinum based chemotherapy, who also subsequently progressed during or after a platinum-doublet regimen given to treat the recurrence, are eligible.
5. Life expectancy ≥ 12 weeks.
6. ECOG performance status of 0 or 1.
7. The main organ's function is normal and it should meet the following criteria:

   Blood routine examination should be complied with (No blood transfusion, no use of hematopoietic factors and no use of drugs for correction within 14 days):
   1. ANC ≥ 1.5×109/L；
   2. PLT ≥ 100×109/L；
   3. HB ≥ 90 g/L；
   4. ALB ≥ 30 g/L
   5. TSH ≤ ULN (however, patients with free Triiodothyronine [FT3] or free Thyroxine [FT4] levels ≤ ULN may be enrolled)
   6. TBIL ≤ULN；
   7. ALT、AST≤ 1.5 ULN
   8. AKP≤2.5 ULN
   9. Cr≤1.5ULN，endogenous creatinine clearance rate≥60ml/min(Cockcroft-Gault formula);
8. Women of childbearing age must undergo a serological pregnancy test within 7 days before the first dose with negative results and willing to use a medically approved and effective contraceptive method (e.g. intrauterine device, contraceptive pill or condom) during the study and within two months after the last dose. For male subjects whose partners are women of childbearing age, they should be sterilized surgically or agree to use effective contraceptive methods during the study and within two months after the last dose.
9. Subjects should be voluntarily participate in clinical studies and informed consent should be signed.

Exclusion Criteria:

1. Subjects have a history of any active autoimmune disease or autoimmune disease including but not limited to the following: autoimmune hepatitis,interstitial pneumonia,uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism which can be included after hormone replacement therapy; Subjects with childhood asthma have been completely alleviated and without any intervention or vitiligo in adulthood can be included. Subjects who need medical intervention with bronchodilators can not be included.
2. Participated in other clinical trials, or finish other clinical trials within 4 weeks.
3. Known history of hypersensitivity to any components of the Camrelizumab formulation，or other monoclonal antibody.
4. Known history of hypersensitivity to paclitaxel or albumin human .
5. Peripheral blood neutrophils <1500/mm3
6. Subjects with epidermal growth factor receptor (EGFR)-sensitizing mutation and/or anaplastic lymphoma kinase (ALK) translocation.
7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least two months prior to the first dose of trial treatment and any Neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 14 days prior to trial treatment.
8. Clinically significant cardiovascular diseases, including but not limited to congestive heart failure (New York heart association (NYHA) class > 2), unstable or severe angina, severe acute myocardial infarction within 1 year before enrollment, supraventricular or ventricular arrhythmia which need medical intervention.
9. Subjects with congenital or acquired immunodeficiency such as HIV infection, active hepatitis B (HBV DNA ≥ 2000 IU/ml), hepatitis C (hepatitis C antibody is positive).
10. Subjects with other factors that might lead to the termination of the study, such as serious diseases (including mental illness) requiring combined treatment, severe laboratory abnormality, and family or social factors，which will affect the safety of the subjects, or the collection of data and samples. in the opinion of the treating Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 12 months
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

SECONDARY OUTCOMES:
12-month PFS rate | From date of enrollment up to 12 months
  The rate of 12-month PFS
Progression-free Survival (PFS) | Time Frame: Up to approximately 24 months
  Progression-free survival is defined as the duration from date of enrollment to the first occurrence of progression of disease or death from any cause
Overall survival (OS) | Up to approximately 24 months
  Overall survival is defined as the duration from date of enrollment to the date of death from any cause.
Duration of Response (DCR) | Up to approximately 24 months
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or stable disease (SD) per RECIST 1.1.
Duration of Response (DOR) | Up to approximately 24 months
  DOR is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Incidence of Adverse Events (AEs) in the treatment of Camrelizumab in combination with nb-Paclitaxel | Up to approximately 24 months
  Number of participants with adverse events occurring up to 30 days after the last administration are evaluated and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03.

OTHER OUTCOMES:
PD-L1 expression on tumor and immune cells | Up to approximately 24 months
  The efficacy of the combination of Camrelizumab and nb-Paclitaxel as measured by objective response, will be described in patients according to PD-L1 positive and PD-L1 negative.
Tumor Mutation Burden (TMB) | Up to approximately 24 months
  The impact of TMB on efficacy of the combination of Camrelizumab and nb-Paclitaxel will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuyu Cai, MD, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The first affiliated hospital of guangzhou medical university, Guangzhou, Guangdong
  - The First Affiliated Hospital/School of Clinical Medicine of Guangdong Pharmaceutical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided
Update after discussion